CLINICAL TRIAL: NCT06747000
Title: Lipoprotein Functions in Healthy Individuals and Subjects With Lipid Disorders
Brief Title: Lipoprotein Interactions and Platelet Function in Healthy Individuals and Those With Lipid Disorders
Status: Recruiting | Type: Observational
Sponsor: The Miriam Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2195890; 710-7149062 (Other Grant/Funding Number: Departmental)
Record Dates: First submitted 2024-12-18; First posted 2024-12-24 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Lipid Disorders
Keywords: lipids; lipoproteins; platelets; high cholesterol
MeSH Terms: conditions — Lipid Metabolism Disorders; Hypercholesterolemia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Individuals with lipid disorders: Individuals with lipid disorders (elevated HDL and LDL)
- Healthy individuals: Healthy individuals with normal lipid values and without lipid-related diseases

SUMMARY:
This study looks at how lipoproteins, which are particles in the blood that transport cholesterol, influence heart and blood vessel health. Beyond just their levels, the way these particles function plays a key role in preventing or contributing to disease. In some conditions, like high cholesterol or diabetes, lipoproteins may not work properly, increasing the risk of clogged arteries and other complications.

The investigators aim to study these changes in people with lipid disorders to better understand their impact on blood health and to find new ways to prevent and treat heart disease.

DETAILED DESCRIPTION:
Traditionally, lipoproteins have been associated with cardiovascular protection, but emerging research indicates that their functionality may be a more critical factor than their levels in evaluating cardiovascular risk. Lipoproteins, such as HDL, LDL, and VLDL, play vital roles in processes like reverse cholesterol transport and demonstrate anti-inflammatory, antioxidative, and antiplatelet properties. However, in conditions like atherosclerosis, diabetes, and dyslipidemia, these lipoproteins often become dysfunctional, and the mechanisms behind this dysfunction remain incompletely understood.

This study aims to thoroughly investigate the pathogenic roles of lipoproteins by examining their structural and functional modifications and their influence on platelet activity in individuals with lipid disorders.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers
* Abnormalities in lipid panels
* Able to provide informed consent
* Between the age of 18 and 69

Exclusion Criteria:

* Drug or alcohol abuse within 6 months or significant mental/psychological impairment
* Current smokers
* Subjects with known bleeding disorders (for example, hemophilia)
* Subjects requiring regular transfusions for any reason
* No ethnic/racial groups will be excluded

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: We Planning to start recruiting process in July 2024. We will identify potential subjects who are seen in the lipid clinic of Lifespan hospitals by EMR review. We will contact potential subjects at a routine care lipid clinic visit or by phone independent of their routine care visits. Recruitment will take place at the Lipid Clinic at Lifespan Hospital, the Brown campus, and our research lab.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2024-07-18 (Actual); Primary Completion 2028-07-18 (Estimated); Study Completion 2029-07-18 (Estimated)

PRIMARY OUTCOMES:
Percentage of platelet aggregation | 5 years
  Platelet aggregation area under the curve will be used as primary endpoint. Specifically, the percentage of platelet aggregation multiple time will be calculated to get area under the curve as a comprehensive marker for platelet aggregation response.

SECONDARY OUTCOMES:
Percentage of Activated Platelets as Assessed by Flow Cytometry | 5 years
  Platelet activation will be assessed as a secondary endpoint. The percentage of activated platelets will be measured using flow cytometry, focusing on markers such as P-selectin expression and fibrinogen binding to the GPIIb/IIIa receptor. Measurements will be taken at multiple time points, and data will be summarized using statistical measures such as mean ± standard deviation.
Plasma levels of CRP in mg/L | 5 years
  Inflammatory markers will be measured as secondary endpoints to evaluate systemic inflammation. Plasma levels of C-reactive protein (CRP) will be reported in milligrams per liter (mg/L) using enzyme-linked immunosorbent assay (ELISA) or similar validated methods. Data will be summarized using statistical measures such as mean ± standard deviation, and comparisons will be made across study groups and time points.
Plasma levels of resolvins in pg/mL | 5 years
  Specialized pro-resolving mediators (SPMs) will be measured as secondary endpoints to assess their role in inflammation resolution. Plasma levels of resolvins will be quantified using liquid chromatography-tandem mass spectrometry (LC-MS/MS) and reported in picograms per milliliter (pg/mL). Data will be summarized using statistical measures such as mean ± standard deviation, and comparisons will be made across study groups and time points.
Plasma Levels of IL-6 in pg/mL | 5 years
  Inflammatory markers will be measured as secondary endpoints to evaluate systemic inflammation. Plasma levels of interleukin-6 (IL-6) will be quantified in picograms per milliliter (pg/mL) using enzyme-linked immunosorbent assay (ELISA) or similar validated methods. Data will be summarized using statistical measures such as mean ± standard deviation, and comparisons will be made across study groups and time points.
Plasma Levels of TNF-α in pg/mL | 5 years
  Inflammatory markers will be measured as secondary endpoints to evaluate systemic inflammation. Plasma levels of tumor necrosis factor-alpha (TNF-α) will be quantified in picograms per milliliter (pg/mL) using enzyme-linked immunosorbent assay (ELISA) or similar validated methods. Data will be summarized using statistical measures such as mean ± standard deviation, and comparisons will be made across study groups and time points.
Plasma levels of protectins in pg/mL | 5 years
  Specialized pro-resolving mediators (SPMs) will be measured as secondary endpoints to assess their role in inflammation resolution. Plasma levels of protectins will be quantified using liquid chromatography-tandem mass spectrometry (LC-MS/MS) and reported in picograms per milliliter (pg/mL). Data will be summarized using statistical measures such as mean ± standard deviation, and comparisons will be made across study groups and time points.
Plasma levels of maresins in pg/mL | 5 years
  Specialized pro-resolving mediators (SPMs) will be measured as secondary endpoints to assess their role in inflammation resolution. Plasma levels of maresins, will be quantified using liquid chromatography-tandem mass spectrometry (LC-MS/MS) and reported in picograms per milliliter (pg/mL). Data will be summarized using statistical measures such as mean ± standard deviation, and comparisons will be made across study groups and time points.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Brown University Health Lipid Clinic, East Providence, Rhode Island
  - Cardiovascular Research Center, Providence, Rhode Island

IPD SHARING:
Plan to Share IPD: Undecided
Currently, the decision regarding sharing IPD has not been finalized. While we recognize the value of data sharing for scientific collaboration, data sharing policies must align with participant confidentiality, regulatory requirements, and institutional policies.